CLINICAL TRIAL: NCT05076006
Title: A Pilot Study to Assess Safety and Biomarker Responses of the Dual JAK1/TYK2 Inhibitor for Cicatricial Alopecia
Brief Title: Dual JAK1/TYK2 Inhibitor for Cicatricial Alopecia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emma Guttman (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Emma Guttman, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 21-0434
Record Dates: First submitted 2021-08-09; First posted 2021-10-13 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Cicatricial Alopecia
Keywords: Alopecia; Scarring Alopecia; Hair Loss
MeSH Terms: conditions — Alopecia | interventions — PF-06700841

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only designated pharmacist will have knowledge of treatment assignment
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Tablets without active ingredients
  Interventions: Drug: Placebo
- PF-06700841 (Experimental): tablets containing active drug (a combined TYK/JAK inhibitor)
  Interventions: Drug: PF-06700841

INTERVENTIONS:
Drug: PF-06700841 — Active study drug
  Other Names: Brepocitinib
  Arms: PF-06700841
Drug: Placebo — placebo comparator
  Arms: Placebo

SUMMARY:
Alopecia could be subdivided into two main groups of diseases: non-scarring alopecia, such as male pattern baldness, or alopecia areata (AA), in which hair follicles are preserved, yet quiescent, and scarring alopecia, also known as cicatricial alopecia (CA), in which hair follicles are irreversibly destroyed. CA leads to scarred areas, most commonly on the scalp, that cannot re-grow hair. Despite being a long-term condition, that often has significant impact on patients' well-being, available effective treatments for these diseases are lacking. In addition, the molecular abnormalities causing CA are largely unknown. The study team's research involves administrating patients a new investigational drug (a combined TYK/JAK inhibitor) which has been shown to be safe and well tolerated in clinical studies to date, and is being investigated in other conditions, such as AA. CA patients will be asked to provide small samples of skin and blood throughout the treatment period, to find out how they respond to the drug, and to attempt to better understand these diseases.

DETAILED DESCRIPTION:
JAK inhibitors are a group of small molecules, recently emerging as an appealing class of immune modifiers in dermatology. These are antagonists of the various members of the JAK enzymes family, which consists of JAK1, JAK2, JAK3, and tyrosine kinase-2 (TYK2). JAKs enable the binding and activation of the transducer and activator of transcription (STAT), by phosphorylating the cytoplasmic domain of multiple cytokine receptors. This results in translocation of the STAT into the nucleus, which greatly affects transcription. JAK antagonism therefore blocks this signaling through STAT activation, targeting Th1/IFN-γ as well as common γc cytokines (shared between IL-2, IL-4, IL-9, IL-7, IL-15 and IL-21), and TYK2 also adds an IL-23 capability. Therefore PF-06700841, a dual inhibitor of JAK1 and TYK2, currently being investigated for a number of indications including psoriasis, Crohn's disease, ulcerative colitis, psoriatic arthritis, atopic dermatitis, psoriasis, systemic lupus erythematosus and AA, and which has been shown to be safe and well tolerated, with good safety profile, was chosen for this protocol.

The study team will evaluate scalp and blood markers of inflammation, hair keratins and fibrosis, and our ultimate goal would be to elucidate the relations between inflammation and tissue scarring. While the study design is specifically powered to detect mechanistic tissue effects of PF-06700841, drug safety and tolerability in this patient population will also be closely monitored.

The study team's research proposal is novel in that the team proposes to investigate the immune profile of CA patients in skin and blood, at baseline, as well as during treatment with PF-06700841. In addition to the much-needed, prospective investigation of a new treatment modality for these diseases, the study team also aims to better characterize these diseases molecularly, and attempt to determine the effects of the inflammatory process on the resultant fibrosis. These findings will help to identify new treatment targets as well as direct further investigation for the development of new therapies for these disfiguring diseases.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of any gender, age 18 years or older, at the time of informed consent at Screening
* Subjects who are willing and able to adhere to the study visit schedule and comply with protocol requirements.
* Subject self-reports active CA (LPP/FFA or CCCA). for at least 6 months from screening visit. Diagnosis will be confirmed clinically at screening visit.
* Subject has a negative Tuberculin purified protein derivative (PPD) or QuantiFERON TB-Gold test (QFT) at screening.
* Subject is judged to be in otherwise good overall health following a detailed medical and medication history, physical examination, and laboratory testing.

Exclusion Criteria:

* Subject's cause of hair loss is indeterminable and/or they have concomitant causes of alopecia, such pregnancy-related, drug-induced, telogen effluvium, or advanced androgenetic alopecia.
* Subject has a history of CA for ≥ 7 years since their disease onset, severe fibrosing disease, or very rapid hair loss.
* Subject has a history of moderate to severe keloids on the scalp, as determined by clinical examination at screening.
* Other scalp disease that may impact assessment (eg, scalp psoriasis, dermatitis, etc).
* Subject is pregnant or breastfeeding. Female subjects of childbearing potential must agree to use two effective methods (one of which is a highly effective method) of contraception throughout the study and for at least 28 days after the last dose of investigational product. Women of childbearing potential must test negative for pregnancy prior to enrollment in this study.
* Participation in other studies involving investigational drug(s) within 8 weeks or within 5 half-lives (if known), whichever is longer, prior to study entry and/or during study participation.
* Active systemic diseases that may cause hair loss (eg, systemic lupus erythematosus, thyroiditis, systemic sclerosis, lichen planus, etc).
* Any Psychiatric condition in the opinion of the investigator precludes participation in the study .
* Current or recent history of clinically significant severe, progressive, or uncontrolled renal (including but not limited to active renal disease or recent kidney stones), hepatic, hematological, gastrointestinal, metabolic, endocrine (particularly thyroid disease which can be associated with hair loss), pulmonary, cardiovascular, psychiatric, immunologic/rheumatologic or neurologic disease; or have any other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration, or interfere with the interpretation of study results; or in the opinion of the investigator, the subject is inappropriate for entry into this study, or unwilling/unable to comply with STUDY PROCEDURES.
* Any present malignancies or history of malignancies with the exception of adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ.
* History of any lymphoproliferative disorder such as Epstein Barr Virus (EBV) related lymphoproliferative disorder, history of lymphoma, history of leukemia, or signs and symptoms suggestive of current lymphatic or lymphoid disease.
* History (single episode) of disseminated herpes zoster or disseminated herpes simplex, or a recurrent (more than one episode of) localized, dermatomal herpes zoster.
* History of systemic infection requiring hospitalization, parenteral antimicrobial therapy, or as otherwise judged clinically significant by the investigator within 6 months prior to Day 0.
* Active acute or chronic infection requiring treatment with oral antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 4 weeks prior to Day 0 or superficial skin infection within 1 week prior to Day 0.
* Significant trauma or major surgery within 1 month of signing informed consent.
* Considered in imminent need for surgery or with elective surgery scheduled to occur during the study.
* Active hepatitis B, hepatitis C, human immunodeficiency virus (HIV), or positive HIV serology at the time of screening for subjects determined by the investigators to be at high-risk for this disease.
* Have an active history of alcohol or substance abuse within 1 year prior to Day 0.
* Donation of blood in excess of 500 mL within 8 weeks prior to Day 0.
* Subject has received a live attenuated vaccine ≤ 30 days prior to study screening.
* Subject has any uncertain or clinically significant laboratory abnormalities that may affect interpretation of study data or endpoints, at determined by the PI.
* History of adverse systemic or allergic reactions to components of study drug.
* Use of systemic immunosuppressive medications, including, but not limited to, cyclosporine, systemic or intralesional corticosteroids, mycophenolate mofetil, azathioprine, methotrexate, within 8 weeks prior to baseline visit.
* Use of other systemic agent for CA, including, 5α-reductase inhibitors, hydroxychloroquine, or retinoids, within 4 weeks prior to baseline visit.
* Use of an intralesional corticosteroids or oral JAK inhibitor (tofacitinib, ruxolitinib) within 4 weeks prior to the baseline visit.
* Subject has used topical corticosteroids, and/or tacrolimus, and/or pimecrolimus within 1 week before the baseline visit.
* Subject has been previously treated with biological drugs in the last 12 weeks for other indications.
* Subjects previously tested with a positive or indeterminable PPD or QFT result, including subjects that completed standard tuberculosis therapy.
* Screening 12-lead ECG that demonstrates clinically significant abnormalities requiring treatment, e.g acute myocardial infarction, serious tachy or brady arrhythmias or that are indicative of serious underlying heart disease (e.g. cardiomyopathy, major congenital heart disease, low voltage in all leads, Wolff-Parkinson-White syndrome and other clinically relevant abnormalities which may affect participant safety or interpretation of study results. A history of additional risk factors for Torsades de Pointes (TdP) (e.g. heart failure, hypokalemia, family history of long QT syndrome).
* If QTcF exceeds 450 mS, or QRS exceeds 120 mS, the ECG should be repeated 2 more times and the average of 3 QTc or QRS values should be used to determine the participants' eligibility. Participants with average screening value QTcF > 450 mS should be excluded. Concomitant use of medications that prolong the QT/QTcF interval is exclusionary.
* Use of concomitant drugs that prolong the QT interval at the judgment of the PI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence and Severity of Treatment-Emergent adverse events | Week 48
  The adverse event will be described and categorized as Treatment-emergent, Serious, abnormal in vital signals, and abnormal in laboratory parameters.
Changes from baseline in CCL5 gene expression level in response to PF-06700841 | Week 12 and Week 24
  mRNA Levels of CCL5 gene expression in skin biopsies quantified by normalized Ct values obtained by quantitative real-time PCR assay, measured at baseline, week 12 and week 24. Changes are characterized by differences in Ct values from a specific time point (week 12 or week 24) to baseline.
Changes from baseline in CXCR3 gene expression level in response to PF-06700841 | Week 12 and Week 24
  mRNA Levels of CXCR3 gene expression in skin biopsies quantified by normalized Ct values obtained by quantitative real-time PCR assay, measured at baseline, week 12 and week 24. Changes are characterized by differences in Ct values from a specific time point (week 12 or week 24) to baseline.

SECONDARY OUTCOMES:
Changes from baseline in IFN-γ gene expression level in response to PF-06700841 | Week 12, Week 24 and Week 48
  mRNA Levels of IFN-γ gene expression in skin biopsies quantified by normalized Ct values obtained by quantitative real-time PCR assay, measured at baseline, week 12, week 24 and week 48. Changes are characterized by differences in Ct values from a specific time point (week 12, week 24 or week 48) to baseline.
Changes from baseline in CXCL9 gene expression level in response to PF-06700841 | Week 12, Week 24 and Week 48
  mRNA Levels of CXCL9 gene expression in skin biopsies quantified by normalized Ct values obtained by quantitative real-time PCR assay, measured at baseline, week 12, week 24 and week 48. Changes are characterized by differences in Ct values from a specific time point (week 12, week 24 or week 48) to baseline.
Changes from baseline in CXCL10 gene expression level in response to PF-06700841 | Week 12, Week 24 and Week 48
  mRNA Levels of CXCL10 gene expression in skin biopsies quantified by normalized Ct values obtained by quantitative real-time PCR assay, measured at baseline, week 12, week 24 and week 48. Changes are characterized by differences in Ct values from a specific time point (week 12, week 24 or week 48) to baseline.
Changes from baseline in IL-12RB1 gene expression level in response to PF-06700841 | Week 12, Week 24 and Week 48
  mRNA Levels of IL-12RB1 gene expression in skin biopsies quantified by normalized Ct values obtained by quantitative real-time PCR assay, measured at baseline, week 12, week 24 and week 48. Changes are characterized by differences in Ct values from a specific time point (week 12, week 24 or week 48) to baseline.
Changes from baseline in STAT1 gene expression level in response to PF-06700841 | Week 12, Week 24 and Week 48
  mRNA Levels of STAT1 gene expression in skin biopsies quantified by normalized Ct values obtained by quantitative real-time PCR assay, measured at baseline, week 12, week 24 and week 48. Changes are characterized by differences in Ct values from a specific time point (week 12, week 24 or week 48) to baseline.
The Frontal Fibrosis Alopecia Severity Index (FFASI) | Baseline
  The Frontal Fibrosis Alopecia Severity Index utilizes clinical images of the entire hairline divided into 4 sections. Score from 1-5, with higher score indicating more severity.
The Frontal Fibrosis Alopecia Severity Index (FFASI) | Week 12
  The Frontal Fibrosis Alopecia Severity Index utilizes clinical images of the entire hairline divided into 4 sections. Score from 1-5, with higher score indicating more severity.
The Frontal Fibrosis Alopecia Severity Index (FFASI) | Week 24
  The Frontal Fibrosis Alopecia Severity Index utilizes clinical images of the entire hairline divided into 4 sections. Score from 1-5, with higher score indicating more severity.
The Frontal Fibrosis Alopecia Severity Index (FFASI) | Week 48
  The Frontal Fibrosis Alopecia Severity Index utilizes clinical images of the entire hairline divided into 4 sections. Score from 1-5, with higher score indicating more severity.
The Lichen Planopilaris Activity Index (LPPAI) | Baseline
  The Lichen Planopilaris Activity Index is a numeric composite index that aggregates symptoms and signs of pruritus, pain, burning, scalp erythema , perifollicular erythema, perifollicular scale , pull test and spreading. Symptoms and signs are measured in a 4-point scale (0-absent, 1-mild, 2-moderate and 3-severe). Full range from 0-10, higher score indicates more severity.
The Lichen Planopilaris Activity Index (LPPAI) | Week 12
  The Lichen Planopilaris Activity Index is a numeric composite index that aggregates symptoms and signs of pruritus, pain, burning, scalp erythema , perifollicular erythema, perifollicular scale , pull test and spreading. Symptoms and signs are measured in a 4-point scale (0-absent, 1-mild, 2-moderate and 3-severe). Full range from 0-10, higher score indicates more severity.
The Lichen Planopilaris Activity Index (LPPAI) | Week 24
  The Lichen Planopilaris Activity Index is a numeric composite index that aggregates symptoms and signs of pruritus, pain, burning, scalp erythema , perifollicular erythema, perifollicular scale , pull test and spreading. Symptoms and signs are measured in a 4-point scale (0-absent, 1-mild, 2-moderate and 3-severe). Full range from 0-10, higher score indicates more severity.
The Lichen Planopilaris Activity Index (LPPAI) | Week 48
  The Lichen Planopilaris Activity Index is a numeric composite index that aggregates symptoms and signs of pruritus, pain, burning, scalp erythema , perifollicular erythema, perifollicular scale , pull test and spreading. Symptoms and signs are measured in a 4-point scale (0-absent, 1-mild, 2-moderate and 3-severe). Full range from 0-10, higher score indicates more severity.
The Central Hair Loss Grade (CHLG) | Baseline
  The Central Hair Loss Grade is a clinical measure of severity that uses a 6 points scale (0 no central scalp hair loss , 1 - minimal central scalp hair loss , 2 - clinically evident central scalp hair loss, 3-5 advanced central scalp hair loss)
The Central Hair Loss Grade (CHLG) | Week 12
  The Central Hair Loss Grade is a clinical measure of severity that uses a 6 points scale (0 no central scalp hair loss , 1 - minimal central scalp hair loss , 2 - clinically evident central scalp hair loss, 3-5 advanced central scalp hair loss)
The Central Hair Loss Grade (CHLG) | Week 24
  The Central Hair Loss Grade is a clinical measure of severity that uses a 6 points scale (0 no central scalp hair loss , 1 - minimal central scalp hair loss , 2 - clinically evident central scalp hair loss, 3-5 advanced central scalp hair loss)
The Central Hair Loss Grade (CHLG) | Week 48
  The Central Hair Loss Grade is a clinical measure of severity that uses a 6 points scale (0 no central scalp hair loss , 1 - minimal central scalp hair loss , 2 - clinically evident central scalp hair loss, 3-5 advanced central scalp hair loss)
Change in Physician Global Assessment of Improvement (PGA-I) | Week 24
  The PGA-I ranges from -4(significant worsening) to 4(significant improvement).
Change in Physician Global Assessment of Improvement (PGA-I) | Week 28
  The PGA-I ranges from -4(significant worsening) to 4(significant improvement).
Change in the Dermatology Quality of Life Index (DLQI) | Baseline
  DLQI is a questionnaire with quality of life indicators related to the health of the skin. This questionnaire has 10 items related to skin problems, each one with 4 possible answers: Very Much, A Lot, A Little, and Not at All. The sum of items scores will generate a score of how much the skin problem affects the personal life. Full score range from 0 to 30, with higher score indicating poorer health outcomes.
Change in the Dermatology Quality of Life Index (DLQI) | Week 12
  DLQI is a questionnaire with quality of life indicators related to the health of the skin. This questionnaire has 10 items related to skin problems, each one with 4 possible answers: Very Much, A Lot, A Little, and Not at All. The sum of items scores will generate a score of how much the skin problem affects the personal life. Full score range from 0 to 30, with higher score indicating poorer health outcomes.
Change in the Dermatology Quality of Life Index (DLQI) | Week 24
  DLQI is a questionnaire with quality of life indicators related to the health of the skin. This questionnaire has 10 items related to skin problems, each one with 4 possible answers: Very Much, A Lot, A Little, and Not at All. The sum of items scores will generate a score of how much the skin problem affects the personal life. Full score range from 0 to 30, with higher score indicating poorer health outcomes.
Change in the Dermatology Quality of Life Index (DLQI) | Week 48
  DLQI is a questionnaire with quality of life indicators related to the health of the skin. This questionnaire has 10 items related to skin problems, each one with 4 possible answers: Very Much, A Lot, A Little, and Not at All. The sum of items scores will generate a score of how much the skin problem affects the personal life. Full score range from 0 to 30, with higher score indicating poorer health outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Guttman, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-05-30): https://cdn.clinicaltrials.gov/large-docs/06/NCT05076006/ICF_000.pdf